CLINICAL TRIAL: NCT07165184
Title: A Prospective Observational Study of Subcarinal Lymph Node Metastasis in Patients With Esophageal Cancer
Brief Title: Incidence of 107 Lymph Node Metastasis
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director, Institute of Thoracic Oncology, Fudan University, Fudan University
Other Study IDs: ECTOP-2009
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer
Keywords: esophagectomy; lymph node metastasis
MeSH Terms: conditions — Esophageal Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group: All patients who had surgery due to esophageal cancer with curative intent, no intervention was applied.
  Interventions: Other: no intervention was applied as observation study

INTERVENTIONS:
Other: no intervention was applied as observation study — no intervention was applied as observation study

SUMMARY:
the study was to document the incidence o subcarinal lymph node metastasis, and the risk factors of metastasis.

DETAILED DESCRIPTION:
Esophageal cancer remains one of the most prevalent malignancies worldwide, with surgery serving as the cornerstone for resectable cases. Although patient survival has improved with the integration of chemotherapy, radiotherapy, and immunotherapy, esophageal surgery still carries a high risk of postoperative complications despite recent technical advancements. Standard procedures involve tumor resection, digestive tract reconstruction, and comprehensive lymphadenectomy.

Our prior research demonstrated that complete right thoracic lymph node dissection significantly enhances long-term survival compared to incomplete left thoracic dissection (1). However, extended three-field dissection offered no survival advantage over conventional two-field dissection (2), necessitating further refinement of the latter's scope. Current preoperative diagnostics for lymph node metastasis suffer from limited sensitivity (3). During traditional two-field dissection, removing subcarinal lymph nodes (located below the carina) may compromise tracheobronchial blood supply, increasing risks of postoperative cough and pneumonia. Our retrospective study revealed a low subcarinal metastasis rate of approximately 2% (4). The risk factors and long-term prognostic impact of subcarinal metastasis remain unclear, requiring prospective studies to validate the necessity of this nodal station dissection.

This prospective study aims to investigate the incidence and risk factors of subcarinal lymph node metastasis within conventional dissection ranges, providing robust evidence for personalized treatment strategies in esophageal cancer.

reference：

1. Li B, Hu H, Zhang Y, et al. Extended Right Thoracic Approach Compared With Limited Left Thoracic Approach for Patients With Middle and Lower Esophageal Squamous Cell Carcinoma: Three-year Survival of a Prospective, Randomized, Open-label Trial. Ann Surg . 2018 May;267(5):826-832.
2. Li B, Zhang Y, Miao L, et al. Esophagectomy With Three-Field Versus Two-Field Lymphadenectomy for Middle and Lower Thoracic Esophageal Cancer: Long-Term Outcomes of a Randomized Clinical Trial. J Thorac Oncol . 2021 Feb;16(2):310-317.
3. Li B, Li N, Liu S, et al. Does [18F] fluorodeoxyglucose-positron emission tomography/computed tomography have a role in cervical nodal staging for esophageal squamous cell carcinoma? J Thorac Cardiovasc Surg . 2020 Aug;160(2):544-550.
4. Lin K, Li B, Sun Y, et al. Precise pattern of lymphatic spread of esophageal squamous cell carcinoma: results of 1074 patients with N1 disease. J Cancer Res Clin Oncol . 2023 Nov;149(17):15819-15825

ELIGIBILITY:
Inclusion Criteria:

* patients with esophageal squamous cell carcinoma
* clinical staging: cT1-4a N0/+ M0.
* no history of other malignancy.

Exclusion Criteria:

* esophageal cancer in the neck
* poor physical status to have esophagectomy.

Ages: 20 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who had surgery due to esophageal cancer with curative intent
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2027-07-21 (Estimated); Study Completion 2030-07-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of left subcarinal lymph node metastasis | 2 years
  number of patients who had subcarinal lymph node metastasis/number of patients who had resection of subcarinal lymph node

SECONDARY OUTCOMES:
Risk factors of subcarinal lymph node metastasis | 2 years
  risk factors that related to the metastasis of subcarinal lymph node.
Survival of patients with subcarinal ymph node metastasis | 3 years
  the disease-free survival and overall survival of patients who had subcarinal lymph node metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
the IPD and supporting information will be available from January 1st 2027 to December 31st 2030.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code